CLINICAL TRIAL: NCT06960759
Title: Mechanisms of Change in Behavioral Cough Suppression Therapy for Refractory Chronic Cough
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Montana (Other)
Collaborators: University of Colorado, Denver (Other); Emory University (Other); University of Melbourne (Other)
Responsible Party: Principal Investigator, Laurie Slovarp, Professor, University of Montana
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 25-0206
Record Dates: First submitted 2025-04-28; First posted 2025-05-07 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Chronic Cough (CC); Refractory Chronic Cough; Unexplained Chronic Cough
Keywords: cough hypersensitivity syndrome; randomized control trial; neurogenic cough; refractory chronic cough; unexplained chronic cough; chronic cough; behavioral cough suppression therapy
MeSH Terms: conditions — Chronic Cough; cough hypersensitivity syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Behavioral treatment plus inactive drug (Active Comparator): Participants receive behavioral cough suppression therapy (BCST) combined with an inactive inhaled substance.
  Interventions: Behavioral: Behavioral cough suppression therapy combined with inactive inhaled drug (BCS+Sham)
- Behavioral treatment plus inhaled drug (Experimental): Participants receive behavioral cough suppression therapy (BCST) combined with inhaled vaporized drug designed to enhance BCST
  Interventions: Combination Product: Behavioral cough suppression therapy combined with capsaicin inhalation (BCS+CAP)
- Inhaled drug (Experimental): Participants inhale a drug designed to desensitize the cough reflex.
  Interventions: Drug: Inhaled capsaicin (CAP)

INTERVENTIONS:
Behavioral: Behavioral cough suppression therapy combined with inactive inhaled drug (BCS+Sham) — Behavioral cough suppression therapy plus inactive inhaled drug. Treatment given twice per week for 12 sessions.
  Arms: Behavioral treatment plus inactive drug
Combination Product: Behavioral cough suppression therapy combined with capsaicin inhalation (BCS+CAP) — Behavioral cough suppression therapy combined with inhaled capsaicin (cough stimulant). Treatment given twice per week for 12 sessions.
  Arms: Behavioral treatment plus inhaled drug
Drug: Inhaled capsaicin (CAP) — Repeated inhalation of diluted capsaicin in increasing concentrations. Treatment given twice per week for 12 sessions.
  Arms: Inhaled drug

SUMMARY:
This study is testing new ways to help people who have chronic cough that has not improved with typical treatments. One approach is called behavioral cough suppression (BCS) therapy, which teaches people techniques to stop themselves from coughing. Another approach uses capsaicin, the substance that makes chili peppers hot, to help reduce the body's sensitivity to cough triggers.

In this study, we will test three treatments:

* BCS therapy with capsaicin (BCS+CAP),
* BCS therapy with a placebo (BCS+Sham),
* Capsaicin stimulation alone (CAP).

The investigators will enroll 150 adults with chronic cough and randomly assign them to one of the three treatments. Each person will attend 12 treatment sessions.

The investigators want to find out how these treatments affect:

* How sensitive someone is to things that make them cough,
* How well they can hold back a cough when they try,
* How their brain responds to things that cause an urge-to-cough,
* And how much their coughing affects their quality of life.

The investigators believe all treatments may reduce sensitivity to cough stimulants, but BCS treatments will also improve how people sense and control the urge to cough. The investigators think combining BCS with capsaicin will work the best overall.

DETAILED DESCRIPTION:
Refractory chronic cough (RCC) is a persistent and costly condition that is difficult to treat, often persisting despite appropriate treatment of underlying causes. While behavioral cough suppression (BCS) therapy has shown effectiveness in reducing cough frequency and improving quality of life in controlled studies, it remains underutilized, and the mechanisms by which it works are not well understood.

This multi-site randomized controlled trial will investigate the effects and mechanisms of BCS therapy with and without the addition of capsaicin desensitization, compared to capsaicin stimulation alone. Capsaicin, a known cough stimulant, has demonstrated desensitization effects on sensory pathways in conditions such as chronic rhinitis and pain syndromes, suggesting potential utility in modulating cough-related neural pathways.

The investigators will recruit 150 participants diagnosed with RCC and randomize them into one of three treatment arms:

* BCS combined with capsaicin stimulation (BCS+CAP),
* BCS combined with sham stimulation (BCS+Sham),
* Capsaicin stimulation alone (CAP).

Participants will undergo 12 treatment sessions over several weeks. The study will evaluate both behavioral and neural markers of treatment response. Primary outcome measures will include:

* Cough sensory threshold (C5): the lowest concentration of citric acid causing five or more coughs,
* Cough suppression ability: the ability to suppress cough when instructed (the difference between the dose of capsaicin causing five or more coughs when trying to suppress cough (CS5) and C5,
* Urge-to-cough (UTC) sensory-motor threshold difference: a measure of how perception of the need to cough relates to actual coughing behavior,
* Blood oxygen level dependent (BOLD) neural responses using whole-brain functional MRI (fMRI) during UTC stimulation.

Secondary outcomes will include patient-reported measures such as the Leicester Cough Questionnaire (LCQ) and objective ambulatory cough frequency monitoring.

The investigators hypothesize that all three treatments will lead to desensitization of cough sensitivity (i.e., increase in C5), but only the BCS-based interventions will alter UTC thresholds, suppression ability, and brain network activity. We further hypothesize that the combination of BCS and capsaicin (BCS+CAP) will provide the greatest therapeutic benefit due to simultaneous peripheral desensitization and central sensory-motor modulation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of refractory or unexplained chronic cough
* Normal chest x-ray within past 2 years, without change in cough symptoms
* If diagnosed with asthma, is it well controlled
* Normal spirometry (or FEV1/FVC of at least 70% if diagnosed with asthma) within two years, without change in symptoms since
* Laryngoscopy or stroboscopy within 2 years without evidence of structural pathology and no change in vocal quality since exam
* Proficient reader/speaker of English
* Willing to take a pregnancy test before enrollment (if applicable)
* Willing to use contraception during the study (if applicable)
* Demonstrates understanding in study procedures and risks in order to consent

Exclusion Criteria:

* Currently a smoker of any substance
* Currently suffering from any signs of an upper respiratory infection (other than cough)
* Hemoptysis (coughing up blood)
* Pulmonary diagnosis other than asthma
* Used an ACE-inhibitor in the past 60 days
* Pregnant or trying to become pregnant
* Any complaints or clinical symptoms of dysphagia
* Live with or work with anyone with chronic cough

The following additional exclusion criteria will apply to participants at University of Colorado:

* Presence of metal implants, devices or fragments in the body
* Claustrophobia

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2029-06-30 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Cough threshold sensory testing (CTT) | From enrollment to 14 weeks following enrollment
  Measure of cough sensitivity using progressive doses of inhaled vaporized citric acid. The dose causing 5 or more coughs (C5) is the endpoint.
Cough suppression threshold testing (CSTT) | From enrollment to 14 weeks following enrollment
  Measure of cough suppression ability using progressive doses of inhaled vaporized citric acid. The dose causing 5 or more coughs when trying to not cough (CS5) is the endpoint.
Urge-to-Cough Sensory Motor Threshold Difference (UTC S-M Thresh Diff) | From enrollment to 14 weeks following enrollment
  A measure of the relationship between sensation of UTC and motor action of coughing. The measure is determined by calculating the difference between first UTC felt during cough threshold testing (Cu) and UTC at the dose of citric acid that causes 2 or more coughs (C2) (i.e., UTC at C2 - UTC at Cu).
Blood oxygen level dependent neural responses (BOLD) | From enrollment to 14 weeks following enrollment
  Whole-brain fMRI performed during inhalation of capsaicin to trigger urge-to-cough. (NOTE: this measure is only required for those enrolling at Univ. of Colorado)

SECONDARY OUTCOMES:
Leicester Cough Questionnaire (LCQ) | From enrollment to 23 weeks following enrollment
  19-item patient-report outcome measure related to the impact of cough on quality of life
Cough frequency | From enrollment to 14 weeks following enrollment
  Ambulatory cough frequency monitoring with a specialized smartwatch, which is worn for 5 days before treatment and 5 days following treatment

CONTACTS AND LOCATIONS:
Overall Officials: Laurie J Slovarp, PhD, Principal Investigator — University of Montana; Marie Jetté, PhD, Principal Investigator — University of Colorado, Denver
Locations (3):
- United States (3):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Emory University, Atlanta, Georgia
  - University of Montana, Missoula, Montana

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Losche D, Furst W, Falk M, Weickert H. [Preparation of a cytostatic-containing bone cement]. Pharmazie. 1987 Feb;42(2):97-9. German. PMID 3602068
- [Background] Moe AAK, Singh N, Dimmock M, Cox K, McGarvey L, Chung KF, McGovern AE, McMahon M, Richards AL, Farrell MJ, Mazzone SB. Brainstem processing of cough sensory inputs in chronic cough hypersensitivity. EBioMedicine. 2024 Feb;100:104976. doi: 10.1016/j.ebiom.2024.104976. Epub 2024 Jan 19. PMID 38244293
- [Background] Slovarp LJ, Reynolds JE, Tolbert S, Campbell S, Welby S, Morkrid P. Cough desensitization treatment for patients with refractory chronic cough: results of a second pilot randomized control trial. BMC Pulm Med. 2023 Apr 28;23(1):148. doi: 10.1186/s12890-023-02423-6. PMID 37118696
- [Background] Slovarp L, Reynolds JE, Bozarth-Dailey E, Popp S, Campbell S, Morkrid P. Cough desensitization treatment: A randomized, sham-controlled pilot trial for patients with refractory chronic cough. Respir Med. 2022 Mar;193:106739. doi: 10.1016/j.rmed.2022.106739. Epub 2022 Jan 15. PMID 35091204
- [Background] Chamberlain SA, Garrod R, Douiri A, Masefield S, Powell P, Bucher C, Pandyan A, Morice AH, Birring SS. The impact of chronic cough: a cross-sectional European survey. Lung. 2015 Jun;193(3):401-8. doi: 10.1007/s00408-015-9701-2. Epub 2015 Mar 19. PMID 25787221